CLINICAL TRIAL: NCT04724148
Title: Impact of Fentanyl Analgesia on the Accuracy of Hepatic Venous Pressure Gradient Measurements in Patients With Portal Hypertension：a Prospective, Multicenter Study
Brief Title: Impact of Fentanyl Analgesia on the Accuracy of HVPG Measurements in Patients With Portal Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Lishui hospital of Zhejiang University (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fentanyl and HVPG
Record Dates: First submitted 2021-01-11; First posted 2021-01-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Pain
Keywords: hepatic venous pressure gradient; fentanyl
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injecting 1~2mg/kg fentanyl intravenously. (Experimental): 1. Measuring HVPG after the preparation of TIPS in patients with portal hypertension;
  2. Measuring HVPG again 5 minutes later after injecting 1~2mg/kg fentanyl intravenously.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — To assess the accuracy of HVPG in TIPS after injecting a dose of 1~2 mg/kg fentanyl.

SUMMARY:
Portal hypertension is a common complication of chronic liver disease and is associated with most clinical consequences of cirrhosis. The most reliable method for assessing portal hypertension is the measurement of the hepatic venous pressure gradient (HVPG). The HVPG is the gold-standard methods for assessing clinically significant portal hypertension and becoming increasingly used clinically. It is useful in the differential diagnosis of portal hypertension and provides a prognostic index in cirrhotic patients. Many patients are painful and reluctant to undergo serial HVPG measurements. But interventionists are reluctant to use analgesics because they always pay more attention to the accuracy of HVPG measurements.Although Adam F. et al concluded that low-dose midazolam sedation is an option for patients undergoing serial hepatic venous pressure measurements (Hepatology 1999), the effects of using opioid analgesics alone on hepatic venous pressure measurements have not yet been defined. The objective of this study was to evaluate the effects of fentanyl on the HVPG.

DETAILED DESCRIPTION:
Portal hypertension is a common complication of chronic liver disease and is associated with most clinical consequences of cirrhosis. The most reliable method for assessing portal hypertension is the measurement of the hepatic venous pressure gradient (HVPG). The HVPG is the gold-standard methods for assessing clinically significant portal hypertension and becoming increasingly used clinically. It is useful in the differential diagnosis of portal hypertension and provides a prognostic index in cirrhotic patients. Many patients are painful and reluctant to undergo serial HVPG measurements. But interventionists are reluctant to use analgesics because they always pay more attention to the accuracy of HVPG measurements. May be since it is difficult to monitor HVPG for anesthesiologist during liver surgery, there are very few and controversial studies on the effects of sedation and analgesics on HVPG. M. Susan Mandell et al concluded that desflurane alters HVPG measurements, whereas propofol did not change it (Anesth Analg 2003). However, Enric Reverter et al considered that deep sedation with propofol and remifentanil adds substantial variability and uncertainty to HVPG measurements (Liver International 2013). Although Adam F. et al concluded that low-dose midazolam sedation is an option for patients undergoing serial hepatic venous pressure measurements (Hepatology 1999), the effects of using opioid analgesics alone on hepatic venous pressure measurements have not yet been defined. The objective of this study was to evaluate the effects of fentanyl on the HVPG measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and portal hypertension undergoing elective TIPS placement
* ASAⅠ~Ⅲ

Exclusion Criteria:

* Patients with portal vein thrombosis and vein-to-vein communications
* Refusal of consent
* Presence of allergy to fentanyl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of HVPG | 1~2 hours
  To assess whether fentanyl would affect the accuracy of hepatic venous pressure gradient measurements in patients with cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, MD, Study Chair — LanZhou University; Xun Li, MD, Study Chair — LanZhou University; Haijun Zhang, MD, Study Director — LanZhou University; Lei Li, MD, Study Director — LanZhou University; Zhongwei Zhao, MD, Principal Investigator — Lishui hospital of Zhejiang University; Jiansong Ji, PHD, Principal Investigator — Lishui hospital of Zhejiang University; Chuan guang Wang, Master, Principal Investigator — Lishui hospital of Zhejiang University; Wei Wu, Principal Investigator — Lishui hospital of Zhejiang University; Lili Yang, Principal Investigator — Lishui hospital of Zhejiang University; Yulan Li, MD, Principal Investigator — LanZhou University; YuJiang Yin, Principal Investigator — LanZhou University; Wei Yang, master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Zi Niu Yu, MD, Principal Investigator — Zhejiang University; Wentao Wu, master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Xujun Yang, master, Principal Investigator — LanZhou University; Shuangxi Li, Principal Investigator — LanZhou University; Fangyu Xu, Principal Investigator — LanZhou University; Weizhong Zhou, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steinlauf AF, Garcia-Tsao G, Zakko MF, Dickey K, Gupta T, Groszmann RJ. Low-dose midazolam sedation: an option for patients undergoing serial hepatic venous pressure measurements. Hepatology. 1999 Apr;29(4):1070-3. doi: 10.1002/hep.510290421. PMID 10094948
- [Background] Reverter E, Blasi A, Abraldes JG, Martinez-Palli G, Seijo S, Turon F, Berzigotti A, Balust J, Bosch J, Garcia-Pagan JC. Impact of deep sedation on the accuracy of hepatic and portal venous pressure measurements in patients with cirrhosis. Liver Int. 2014 Jan;34(1):16-25. doi: 10.1111/liv.12229. Epub 2013 Jun 13. PMID 23763484
- [Background] Mandell MS, Durham J, Kumpe D, Trotter JF, Everson GT, Niemann CU. The effects of desflurane and propofol on portosystemic pressure in patients with portal hypertension. Anesth Analg. 2003 Dec;97(6):1573-1577. doi: 10.1213/01.ANE.0000090741.63156.1B. PMID 14633521
- [Background] Chinese Portal Hypertension Diagnosis and Monitoring Study Group (CHESS); Minimally Invasive Intervention Collaborative Group, Chinese Society of Gastroenterology; Emergency Intervention Committee, Chinese College of Interventionalists; Hepatobiliary Diseases Collaborative Group, Chinese Society of Gastroenterology; Spleen and Portal Hypertension Group, Chinese Society of Surgery; Fatty Liver and Alcoholic Liver Disease Group, Chineses Society of Hepatology; Chinese Research Hospital Association for the Study of the Liver; Hepatobiliary and Pancreatic Diseases Prevention and Control Committee, Chinese Preventive Medicine Association; Chinese Society of Digital Medicine; Chinese Society of Clinical Epidemiology and Evidence Based Medicine. [Consensus on clinical application of hepatic venous pressure gradient in China (2018)]. Zhonghua Gan Zang Bing Za Zhi. 2018 Nov 20;26(11):801-812. doi: 10.3760/cma.j.issn.1007-3418.2018.11.001. No abstract available. Chinese. PMID 30616313
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Qi X, An W, Liu F, Qi R, Wang L, Liu Y, Liu C, Xiang Y, Hui J, Liu Z, Qi X, Liu C, Peng B, Ding H, Yang Y, He X, Hou J, Tian J, Li Z. Virtual Hepatic Venous Pressure Gradient with CT Angiography (CHESS 1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension. Radiology. 2019 Feb;290(2):370-377. doi: 10.1148/radiol.2018180425. Epub 2018 Nov 20. PMID 30457484